CLINICAL TRIAL: NCT05377190
Title: Continuum: Digital Health as Part of the Care Trajectory of Heart Failure Outpatients
Brief Title: Continuum: Digital Health to Manage Heart Failure Outpatients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre hospitalier de l'Université de Montréal (CHUM) (Other)
Collaborators: Greybox (Unknown); Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 2022-10426
Record Dates: First submitted 2022-05-05; First posted 2022-05-17 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2024-08

CONDITIONS: Heart Failure; Chronic Heart Failure
Keywords: Digital health; Digital therapeutics; Software as medical device; Remote patient management; Telemonitoring; Mobile health; Guideline-Directed Medical Therapy
MeSH Terms: conditions — Heart Failure | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- For patients followed in a heart failure clinic (HFC), intervention HFC-IN (Experimental): Use of the full Continuum solution: remote patient monitoring and digital therapeutics over a period of 12 weeks
  Interventions: Other: Continuum HFC-IN
- For patients followed in a HFC, control HFC-IN (Placebo Comparator): Standard of care for the follow-up, no use of remote monitoring or digital therapeutics for the first 12 weeks. After 12 weeks, option is given to the patient to use the full Continuum solution for another period of 12 weeks.
  Interventions: Other: Standard of care for the follow-up
- For patients not followed in a HFC, intervention HFC-OUT (Experimental): Use of part of the Continuum solution: the patient will use a mobile application to enter her/his data but no remote monitoring is performed. Digital therapeutics are used for the healthcare professionals.
  Interventions: Other: Continuum HFC-OUT
- For patients not followed in a HFC, control HFC-OUT (Placebo Comparator): Standard of care for the follow-up, no use of a mobile application or digital therapeutics for the first 12 weeks. After 12 weeks, option is given to the patient to use the mobile app and digital therapeutics are activated for another period of 12 weeks.
  Interventions: Other: Standard of care for the follow-up

INTERVENTIONS:
Other: Continuum HFC-IN — Combination of a mobile application (with remote monitoring) and digital therapeutics
  Arms: For patients followed in a heart failure clinic (HFC), intervention HFC-IN
Other: Standard of care for the follow-up — No mobile application or digital therapeutics are used
  Arms: For patients followed in a HFC, control HFC-IN; For patients not followed in a HFC, control HFC-OUT
Other: Continuum HFC-OUT — Combination of a mobile application (without remote monitoring) and digital therapeutics
  Arms: For patients not followed in a HFC, intervention HFC-OUT

SUMMARY:
Heart failure (HF) is one of the leading causes of hospitalization and death worldwide. Remote patient monitoring and digital therapeutics could help reduce the consumption of care for these patients (hospitalizations, emergency room visits) and optimize their management (education, medication optimization). This randomized study aims to evaluate the effects of the Continuum software solution in patients with heart failure, whether or not they are followed in specialized clinics. Heart failure is one of the main causes of hospitalization and death in the world. Evidence suggests that remote patient monitoring (RPM) and digital therapeutics (DTX solutions) can help improve care consumption (i.e. hospitalizations, emergency visits) and also support health care professionals to improve care (i.e. symptoms management, drug optimization). This randomised study aims to evaluate the effects of these two software solutions in the context of specialized HF clinics (HFC) and primary health care on health care consumption and clinical events.

DETAILED DESCRIPTION:
According to Canadian recommendations, patients recently diagnosed with heart failure or with a recent hospitalization should have a medical follow-up every two to four weeks in order to optimize their treatment and quickly stabilize their condition. However, despite a network of specialized heart failure clinics in the province of Quebec, access to this service is still a challenge because of limited human resources and unequal geographic distribution. Only the most severely ill and unstable patients are followed in these clinics.

The Continuum project combines a remote patient monitoring solution with therapeutic interventions driven by a software to manage heart failure (also called digital therapeutics (DTx)). The patient can send her/his clinical data to the healthcare professional using a mobile application. Healthcare professionals receive not only these data in realtime with potential alerts but also a summarized report of these data and suggested therapeutic interventions.

Our hypotheses are that the Continuum solution, by combining RPM and DTx will 1) improve the workflow and the care trajectory of patients in heart failure clinics resulting in a reduction of cost per patient followed and 2) accelerate drug optimization so they can fully benefit from the recommended therapies for their specific condition.

The general objective of this project is to assess in outpatients the effectiveness of the Continuum solution to reduce healthcare costs and to support medication optimization over a period of 12 weeks.

ELIGIBILITY:
HFC-IN

Inclusion Criteria:

* HF diagnostic
* NYHA 2 or +
* Active follow-up in heart failure clinic
* Ability to use mobile app (or with caregiver's help)
* And one of the following
* New HF diagnosis (<3 months)
* Emergency visit or recent hospitalization with decompensated HF (<6months)
* Increase of >50% diuretic dose, new diuretic or IV diuretic (last 3 months)
* Active heart failure follow-up 2 times in the last 3 months

HFC-OUT

Inclusion Criteria:

* HF diagnostic
* Ability to use mobile app (or with caregiver's help)
* No active follow-up in heart failure clinic or in the waiting list of one

Exclusion Criteria for HFC-IN and HFC-OUT:

* Active hospitalization at randomization or anticipated in the next 2 weeks
* Incapable or minor patient
* History of non-adherence or treatment refusal
* Alcohol or drugs abuse
* Active major depression without caregiver
* Global prognosis < 3months
* Active dialysis or on waiting list
* Heart transplant or mechanical heart
* Severe pulmonary disease with oxygen use or pulmonary transplant waiting list or recurrent pleural drainage
* Severe chronic cirrhosis or hepatic transplant waiting list or recurrent ascites drainage
* Percutaneous or surgical intervention in last 30 days or planned in next 3 months
* Pregnancy
* Active follow-up in another study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 175 (Actual)
Dates: Start 2022-06-08 (Actual); Primary Completion 2023-10-24 (Actual); Study Completion 2023-10-24 (Actual)

PRIMARY OUTCOMES:
CLIC IN ONLY: care consumption | 12 weeks
  Cost analysis on number of hospital (planned or unplanned) ambulatory visits, emergency visits, consultations and hospitalizations
CLIC OUT ONLY: Change in guideline-directed medical therapy by classes | 12 weeks
  Change in guideline-directed medical Therapy optimization between groups before and after intervention by medication classes.
CLIC OUT ONLY: Change in guideline-directed medical therapy by dose | 12 weeks
  Change in guideline-Directed Medical Therapy optimization between groups before and after intervention by medication doses.

SECONDARY OUTCOMES:
CLIC OUT ONLY: Care consumption | 12 weeks
  Cost analysis on number of hospital (planned or unplanned) ambulatory visits, emergency visits, consultations and hospitalizations during intervention
CLIC IN ONLY: Change in guideline-directed medical therapy by classes | 12 weeks
  Compare guideline-Directed Medical Therapy optimization between groups before and after intervention by medication classes
CLIC IN ONLY: Change in guideline-directed medical therapy by doses | 12 weeks
  Compare guideline-Directed Medical Therapy optimization between groups before and after intervention by medication doses
MACE and other clinical events | 12 weeks
  Differences before-after between groups in number of main clinical events including unplanned appointments, emergency consults, all-cause or heart-failure hospitalizations, deaths
CLIC IN ONLY: Quality of life assessment (QoL) with the Kansas City Cardiomyopathy Questionnaire | 12 weeks
  Differences in score before and after
Quality of life assessment (QoL) with the EQ-5D-5L EuroQOL instrument | 12 weeks
  Differences in score before and after
New York Heart Association class | 12 weeks
  A reduction of at least one class in New York Heart Association (NYHA) scale
NTproBNP | 12 weeks
  Reduction in NTproBNP greater than 30%
Pharmacological profile | 12 weeks
  Percentage of recommended heart failure drugs prescribed

CONTACTS AND LOCATIONS:
Overall Officials: François Tournoux, MD PhD, Principal Investigator — CHUM
Locations (1):
- CRCHUM, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Marier-Tetrault E, Bebawi E, Bechard S, Brouillard P, Zuchinali P, Remillard E, Carrier Z, Jean-Charles L, Nguyen JNK, Lehoux P, Pomey MP, Ribeiro PAB, Tournoux F. Remote Patient Monitoring and Digital Therapeutics Enhancing the Continuum of Care in Heart Failure: Nonrandomized Pilot Study. JMIR Form Res. 2024 Nov 6;8:e53444. doi: 10.2196/53444. PMID 39504548